CLINICAL TRIAL: NCT00811863
Title: A Prospective Study for the Detection of Nephrogenic Systemic Fibrosis in Patients With Renal Impairment Undergoing Gadoversetamide-enhanced Magnetic Resonance Imaging
Brief Title: Evaluation of Nephrogenic Systemic Fibrosis (NSF) in Patients With Chronic Kidney Disease Following OptiMARK Injection
Acronym: SHERLOC
Status: Withdrawn | Type: Observational
Why Stopped: Study drug currently unavailable
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Other Study IDs: 1177-07-868
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Nephrogenic Systemic Fibrosis; Renal Insufficiency
Keywords: Nephrogenic Systemic Fibrosis; Renal Insufficiency; Gadoversetamide; OptiMARK; Magnetic Resonance Imaging
MeSH Terms: conditions — Nephrogenic Fibrosing Dermopathy; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum; Plasma; Fixed tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Subjects with moderate renal insufficiency defined as an eGFR 30-60 mL/min/1.73 m2
- 2: Subjects with severe renal insufficiency defined as an eGFR <30 mL/min/1.73 m2 and ESRD defined as requiring dialysis

SUMMARY:
The objective of this study is to prospectively monitor the incidence of adverse drug reactions, specifically NSF during routine use of gadoversetamide in a large number of patients with moderate renal insufficiency (eGFR 30-59) and severe renal insufficiency or end-stage renal disease requiring dialysis (eGFR <30).

ELIGIBILITY:
Inclusion Criteria:

* Referred for contrast-enhanced MRI using gadoversetamide;
* Have a documented estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73 m2 within the past 6 months or ESRD requiring dialysis; and
* Willing and able to provide written consent (themselves or by a legally authorized representative) and agree to abide by study requirements, including being seen by a dermatologist and undergoing a skin biopsy if NSF is suspected.

Exclusion Criteria:

* Have experienced a previous hypersensitivity reaction to a GBCA;
* Have pre-existing NSF or NSF-like symptoms; or
* Have been exposed to a GBCA within 12 months prior to the index procedure; or
* Has a medical condition or other personal situation that would prevent providing follow-up information, completing clinic visits or otherwise supplying meaningful data to meet study objectives.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with moderate to severe renal insufficiency that have been identified as requiring (for any indication) a contrast-enhanced MRI using gadoversetamide.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2012-05-17 (Actual); Study Completion 2012-05-17 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the diagnosis of NSF based on clinical assessments and patient telephone calls through 24 months of follow-up. | 1, 3, 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Herbert R. Neuman, MD, Study Director — Mallinckrodt
Locations (1):
- Radiology Consultants, Inc., Youngstown, Ohio, United States